CLINICAL TRIAL: NCT00483093
Title: NGR004:A Phase IB Study of NGR-hTNF in Combination With Cisplatin in Patient Affected by Advanced or Metastatic Solid Tumor
Brief Title: Study of NGR-hTNF in Combination With Cisplatin in Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AGC Biologics S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGR004; 2006-006035-42 (EudraCT Number)
Record Dates: First submitted 2007-06-05; First posted 2007-06-06 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Solid Tumors
Keywords: NGR-hTNF; cisplatin; solid tumors
MeSH Terms: interventions — tumor necrosis factor-alpha, CNGRC fusion protein, human; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: NGR-hTNF; Drug: Cisplatin

INTERVENTIONS:
Drug: NGR-hTNF — iv q3W escalating dose NGR-hTNF up to 1.6 mcg/sqm
Drug: Cisplatin — iv q3W 80 mg/sqm 30 minutes after NGR-hTNF infusion for a maximum of six cycles

SUMMARY:
The main objective of the trial is to document the safety of the combination (escalation doses of NGR-hTNF, from 0.2 mcg/sqm to 1.6 mcg/sqm , with a fixed dose of cisplatin, 80 mg/sqm). Safety will be established by clinical and laboratory assessment according to National Cancer Institute Common Toxicity Criteria (NCI-CTC ).

DETAILED DESCRIPTION:
This is a phase IB, open-label, non-randomized, dose-escalation study that will be conducted in sequential cohorts of patients. Three patients per each cohort are planned.

Patients, with advanced or metastatic solid tumor not amenable of standard therapy will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years with advanced or metastatic solid tumor not amenable to any clinical improvement by current standard treatments and suitable for a treatment with cisplatin

  * Life expectancy more than 3 months
  * ECOG Performance status 0-1
  * Absence of any conditions in which hypervolemia and its consequences (e.g. increased stroke volume, elevated blood pressure) may represent a risk for the patient
  * Adequate baseline bone marrow, hepatic and renal function, defined as follows:
  * Neutrophils > 1.5 x 10^9/L and platelets > 100 x 10^9/L
  * Bilirubin < 1.5 x ULN
  * AST and/or ALT < 2.5 x ULN in absence of liver metastasis
  * AST and/or ALT < 5 x ULN in presence of liver metastasis
  * Serum creatinine < 1.5 x ULN
  * Creatinine clearance (estimated according to Cockcroft-Gault formula) ≥ 50 ml/min
  * Patients may have had prior therapy providing the following conditions are met:
* Chemotherapy, radiation therapy, hormonal therapy or immunotherapy: wash-out period of 28 days
* Corticosteroid therapy wash out period of 14 days
* Surgery: wash-out period of 14 days
* Patients must give written informed consent to participate in the study

Exclusion Criteria:

* Previous signs of severe toxicity platinum related
* Patients must not receive any other investigational agents while on study
* New York Heart Association class III or IV cardiac disease
* Unstable angina
* Patients with myocardial infarction within the last six (6) months
* Patient with significant peripheral vascular disease
* Clinical signs of CNS involvement
* Patients with active or uncontrolled systemic disease/infections or with serious illness or medical conditions, which is incompatible with the protocol
* Known hypersensitivity/allergic reaction to human albumin preparations or to any of the excipients
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol
* Pregnancy or lactation. Patients - both males and females - with reproductive potential (i.e. menopausal for less than 1-year and not surgically sterilized) must practice effective contraceptive measures throughout the study. Women of childbearing potential must provide a negative pregnancy test (serum or urine) within 14 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-07; Primary Completion 2010-06 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
To verify the safety of escalating doses of NGRhTNF (from 0.2 to 1.6 µg/m^2) in combination with cisplatin (80 mg/m^2) every 3 weeks | To recommend a dose regimen of NGR-hTNF + Cisplatin for future phase II trials

SECONDARY OUTCOMES:
To document the preliminary antitumor activity of the combination in terms of objective response rate according to RECIST criteria | every six weeks
To evaluate the pharmacokinetic profiles of the combination of NGR-hTNF and cisplatin | During the study
To measure plasma levels of sTNFRs and anti-NGR-hTNF antibodies | During the study

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Lambaise, MD, Study Director — AGC Biologics S.p.A.
Locations (2):
- Italy (2):
  - Fondazione San Raffaele del Monte Tabor, Milan, Milan,
  - Istituto Europeo Oncologico, Milan, Milan

REFERENCES:
- [Result] Gregorc V, De Braud FG, De Pas TM, Scalamogna R, Citterio G, Milani A, Boselli S, Catania C, Donadoni G, Rossoni G, Ghio D, Spitaleri G, Ammannati C, Colombi S, Caligaris-Cappio F, Lambiase A, Bordignon C. Phase I study of NGR-hTNF, a selective vascular targeting agent, in combination with cisplatin in refractory solid tumors. Clin Cancer Res. 2011 Apr 1;17(7):1964-72. doi: 10.1158/1078-0432.CCR-10-1376. Epub 2011 Feb 9. PMID 21307147